CLINICAL TRIAL: NCT04059458
Title: Biphasic Calcium Phosphate and a Collagen Membrane or Biphasic Calcium Phosphate and Enamel Matrix Proteins, in the Regenerative Treatment of Furcation Grade III Defects
Brief Title: Mandibular Furcation III Regeneration (FURC-III-REGEN)
Acronym: FURC-III-REGEN
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Recruitment problem
Sponsor: University of Oslo (Other)
Responsible Party: Principal Investigator, Anders Verket, Associate Professor, University of Oslo
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FURC-III-REGEN
Record Dates: First submitted 2019-08-06; First posted 2019-08-16 (Actual); Last update posted 2023-11-30 (Actual); Status verified 2023-11

CONDITIONS: Furcation Defects; Periodontal Diseases
MeSH Terms: conditions — Furcation Defects; Periodontal Diseases | interventions — hydroxyapatite-beta tricalcium phosphate; enamel matrix proteins

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Regenerative therapy w/BCP and collagen membrane (Experimental): In this arm, treatment of furcation grade II defects includes open flap debridement and regenerative therapy with biphasic calcium phosphate (BCP) and collagen membrane.
  Interventions: Device: Biphasic calcium phosphate (Straumann Bone Ceramic) + collagen membrane (Straumann Jason Membrane); Drug: Biphasic calcium phosphate (Straumann Bone Ceramic) + enamel matrix proteins (Straumann Emdogain)
- Regenerative therapy w/BCP and enamel matrix proteins (Active Comparator): In this arm, treatment of furcation grade II defects includes open flap debridement and regenerative therapy with biphasic calcium phosphate (BCP) and enamel matrix proteins.
  Interventions: Device: Biphasic calcium phosphate (Straumann Bone Ceramic) + collagen membrane (Straumann Jason Membrane); Drug: Biphasic calcium phosphate (Straumann Bone Ceramic) + enamel matrix proteins (Straumann Emdogain)

INTERVENTIONS:
Device: Biphasic calcium phosphate (Straumann Bone Ceramic) + collagen membrane (Straumann Jason Membrane) — Device: Biphasic calcium phosphate (Straumann Bone Ceramic) + collagen membrane (Straumann Jason Membrane) Following open flap debridement of mandibular grade II furcation defects, regenerative therapy is performed with biphasic calcium phosphate + collagen membrane.
Drug: Biphasic calcium phosphate (Straumann Bone Ceramic) + enamel matrix proteins (Straumann Emdogain) — Drug: Biphasic calcium phosphate (Straumann Bone Ceramic) + enamel matrix proteins (Straumann Emdogain) Following open flap debridement of mandibular grade II furcation defects, regenerative therapy is performed with biphasic calcium phosphate + enamel matrix proteins.

SUMMARY:
Teeth with furcation grade III defects will be treated with open flap debridement and regenerative therapy with biphasic calcium phosphate combined with either enamel matrix proteins or a collagen membrane.

ELIGIBILITY:
Inclusion Criteria:

* Subject must be ≥ 20 years
* Subject must have periodontal disease as determined by the World Workshop 2017 criteria
* Subjects must be undergoing periodontal treatment or follow-up and present 1 or more pair of bilateral mandibular molars affected by furcation involvement grade II with PPD >4 mm, and the furcation fornix must be below a tangential line from the distal to mesial interproximal crestal bone level
* Competent to give consent

Exclusion Criteria:

The following must not be present at the time of enrolment;

* Previous radiotherapy to the jaws, current use of chemotherapy, systemic long-term corticosteroid treatment
* Present or past use of bisphosphonate treatment
* Pregnant or nursing subjects
* Patients classified as > class 2 according to the ASA (American Society of Anesthesiologists) physical status classification
* Previous surgical therapy of included furcation defects
* Inability to comprehend and respond to the quality of life questionnaire
* Dental restorations or prosthesis involving the furcation area
* Root fractures or suspected infractions
* Caries lesions in the furcation area
* No systemic antibiotic treatment within 3 months prior to intervention

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2019-10-15 (Actual); Primary Completion 2023-11-27 (Actual); Study Completion 2023-11-27 (Actual)

PRIMARY OUTCOMES:
Change of furcation grade level | 12 months after treatment
  Proportion of sites demonstrating improvement in furcation grade level as measured with Nabers probe
Change of furcation grade level | 24 months after treatment
  Proportion of sites demonstrating improvement in furcation grade level as measured with Nabers probe

SECONDARY OUTCOMES:
Changes in patient-reported quality of life (QoL) | Preoperatively compared to 24 months after treatment
  To assess QoL changes related to mouth and teeth prior to therapy to after therapy by the use of "The Oral Impacts on Daily Performance (OIDP)" instrument. Each question is assessed by a 5-point scale; (1) never affected, (2) less than once a month, (3) once or twice a month, (4) once or twice a week; and (5) every or nearly every day. The higher number represents more severe impact on quality of life; e.g. worse outcome.
  Each item will be dichotomised yielding the categories (A) affected; including scale categories (2)-(5), and (B) unaffected, including category (1).
Changes in patient-reported quality of life (QoL) | Preoperatively compared to 12 months after treatment
  To assess QoL changes related to mouth and teeth prior to therapy to after therapy by the use of "The Oral Impacts on Daily Performance (OIDP)" instrument. Each question is assessed by a 5-point scale; (1) never affected, (2) less than once a month, (3) once or twice a month, (4) once or twice a week; and (5) every or nearly every day. The higher number represents more severe impact on quality of life; e.g. worse outcome.
  Each item will be dichotomised yielding the categories (A) affected; including scale categories (2)-(5), and (B) unaffected, including category (1).
Changes in defect morphology assessed by CBCT | 24 months after treatment
  Cone beam computed tomography will be acquired at baseline, 2 weeks postoperatively and 24 months postoperatively. This outcome measures quantitative morphologic changes in the furcation defects at 24 months
Changes in pocket probing depth | 12 months after treatment
  Changes in pocket probing depth will be measured with a probe
Changes in pocket probing depth | 24 months after treatment
  Changes in pocket probing depth will be measured with a probe
Changes in PPD | 12 months after treatment
  Changes in pocket probing depth will be measured with a probe
Changes in PPD | 24 months after treatment
  Changes in pocket probing depth will be measured with a probe
Radiographic changes | 12 months after treatment
  Standardized intraoral bitewing radiographs will be obtained and compared to baseline radiographs
Radiographic changes | 24 months after treatment
  Standardized intraoral bitewing radiographs will be obtained and compared to baseline radiographs
Pain following surgery | Up to 1 week postoperatively
  Pain sensation one week posteoperatively will be recorded on a visual analog scale from 0-10. 0 means no pain sensation, whereas 10 means highest pain imagineable.
Caries assessment | 24 months
  Caries in furcation defect assessed with an explorer will be recorded as (Y/N)
Caries assessment | 12 months
  Caries in furcation defect assessed with an explorer will be recorded as (Y/N)

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Clinical Dentistry, Faculty of Dentistry, University of Oslo, Oslo, Norway

IPD SHARING:
Plan to Share IPD: Undecided